CLINICAL TRIAL: NCT02356978
Title: Trial of a New Phototherapy Device for Treating Hyperbilirubinemia in Crigler-Najjar Patients : a New Concept
Brief Title: New Phototherapy Device to Treat Patients With Crigler-Najjar Disease
Acronym: DRAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P140202
Record Dates: First submitted 2015-02-02; First posted 2015-02-06 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2016-12

CONDITIONS: Crigler Najjar Syndrome; Children
Keywords: Rare disease; Crigler-Najjar disease; Paediatric; Experimental device
MeSH Terms: conditions — Crigler-Najjar Syndrome; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Each patient will be treated before using the active usual homemade device, and after using the experimental new "DRAP" device.
  This new sheet was designed by weaving optical fibers connected to LEDs ( "BROCHIER" Technology). The "LIGHTEX" technology ® is a principle of weaving mill of optical fibres with side lighting connected to LEDs and allowing to realize flexible or stiff bright surfaces with very weak congestions, low consumption and high life cycle. The energy illumination of this device varies between 3 and 4 mW / cm ² ( average 3,6 mW / cm ².)
  Interventions: Device: Arm1 homemade phototherapy treatment; Device: DRAP

INTERVENTIONS:
Device: Arm1 homemade phototherapy treatment — session of 10 or 12 hours phototherapy treatment using the homemade device during the first night and then the "DRAP" device during the next nights.
Device: DRAP

SUMMARY:
Evaluating the efficacity of a new device phototherapy by comparing it with conventional phototherapy. Jaundice occurs in many newborns, and is, in most cases benign, However, owing to the potential neurotoxicity of unconjugated bilirubin, newborns must be monitored to identify those who might develop severe hyperbilirubinemia an, in rare cases, acute bilirubin encephalopathy or kernicterus. Treatment of jaundice in newborn relies on phototherapy, exposing their skin to light of a specific wavelength . Fluorescent tubes or halogen lamps have been used as light sources for phototherapy for many years. Light-emitting diodes (LEDs) are more recent sources which are power efficient, have a longer life and are portable with low heat production. Several technologies and devices are developed using LEDs and specially a compact system.

DETAILED DESCRIPTION:
Crigler-Najjar (CN) syndrome is a congenital inborn error of hepatic bilirubin metabolism caused by the deficiency of bilirubin uridinediphosphate glucuronosyltransferase activity CN patients are at permanent risk of life-threatening bilirubin encephalopathy (kernicterus). Treatment of CN disease relies on daily prolonged phototherapy (10-12 h/day). To date, liver transplantation is the only curative treatment available. To date, no phototherapy device exists for teenagers and adults. CN patients use homemade systems or add several neonatal systems together to reach a better efficacy.

A new device has been designed by weaving optical fibers into a sheet connected to LEDs. This new technology, marketed by several manufacturers of phototherapy devices, is used in pediatric wards for treating jaundiced newborns. A prototype of 80× 100cm was thus developed, which combines numerous advantages : important surface of treatment, easy use and transportation, user-friendliness.

Before going to a therapeutic trial for assessing the benefits of this new device in ambulatory current practice, it is essential to make sure of both its feasibility and efficiency on the control of bilirubinemia, under medical supervision.

Hypothesis: the new phototherapy sheet is as effective as, and better tolerated than the usual devices used in CN patients.

ELIGIBILITY:
Inclusion Criteria:

* genetic diagnosis of Crigler Najjar disease
* child whose height is between 60cm and 100cm
* patients with follow-up in reference center,

Exclusion Criteria:

* opposition of parents
* no social security insurance

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Kinetic of blood Bilirubin level using the "DRAP" device (blood bilirubin concentration) | Before using "DRAP" device (H0), and after using (Hour12, Hour 36, Hour 48, Hour 60, Hour 72, Hour 84, Hour 96)
  blood bilirubin concentration will be measured 2 times during phototherapy treatment (before and after phototherapy)

CONTACTS AND LOCATIONS:
Overall Officials: VINCENT GAJDOS, Professor, Principal Investigator — AP-HP, Antoine Béclère Hospital
Locations (1):
- AP-HP, Antoine Béclère Hospital, Clamart, France